CLINICAL TRIAL: NCT00879164
Title: Pilot Evaluation of a Stellate Ganglion Block for the Treatment of Hot Flashes
Brief Title: Stellate Ganglion Nerve Block in Treating Women With Hot Flashes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CDR0000640197; P30CA015083 (NIH); MC08C8 (Other: Mayo Clinic Cancer Center); 08-006796 (Other: Mayo Clinic IRB); NCI-2009-01133 (Other: NCI-CTRP)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Hot Flashes
Keywords: hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bupivacaine hydrochloride
Other: questionnaire administration

SUMMARY:
RATIONALE: A stellate ganglion nerve block may help relieve hot flashes in women.

PURPOSE: This clinical trial is studying how well a stellate ganglion nerve block works in treating women with hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the impact of stellate ganglion blockade on hot flash scores.
* To evaluate the toxicity of stellate ganglion blockade.

OUTLINE: Patients undergo fluoroscopic-guided stellate ganglion blockade using bupivacaine hydrochloride in week 1.

Patients complete a hot flash diary daily and a symptom experience diary weekly in weeks 1-7 and the Profile of Mood States questionnaire in weeks 1 and 7.

After completion of study treatment, patients are followed at 2 months and then monthly for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Presence of hot flashes for ≥ 1 month prior to study registration

  * Hot flashes considered bothersome (defined by their occurrence of ≥ 28 times per week and of sufficient severity to make the patient desire therapeutic intervention)
* Use of more conventional hot flash treatments (including newer antidepressants and gabapentin) have failed to control hot flashes (as defined by the patient)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* Not of childbearing potential, as judged by the attending clinician
* Able to complete questionnaires alone or with assistance
* No evidence of an active malignancy
* No von Willebrand's disease or other bleeding disorders
* No allergy to chlorhexidine or bupivacaine

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior and no concurrent antineoplastic chemotherapy, androgens, estrogens, or progestational agents

  * Tamoxifen, raloxifene, or aromatase inhibitors allowed provided the patient has been on a constant dose for ≥ 4 weeks and continues to receive medication during study treatment
* More than 10 days since prior and no concurrent anticoagulants (e.g., aspirin, clopidogrel, ticlopidine, or warfarin)

  * Concurrent heparin flushes for venous catheter allowed
* No concurrent use of other agents (e.g., megestrol acetate, soy, clonidine, or Bellergal) for treating hot flashes

  * Vitamin E, gabapentin, or antidepressants allowed provided the patient has been on a stable dose for > 30 days and continues to receive medication during study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Difference in hot flash activity between baseline and week 7

SECONDARY OUTCOMES:
Difference in quality of life, toxicity, and self-assessment items between baseline and week 7

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Pachman DR, Barton D, Carns PE, Novotny PJ, Wolf S, Linquist B, Kohli S, Smith DR, Loprinzi CL. Pilot evaluation of a stellate ganglion block for the treatment of hot flashes. Support Care Cancer. 2011 Jul;19(7):941-7. doi: 10.1007/s00520-010-0907-9. Epub 2010 May 23. PMID 20496155